CLINICAL TRIAL: NCT02378467
Title: Saline Hypertonic in Preschoolers
Acronym: SHIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington, the Collaborative Health Studies Coordinating Center (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHIP001
Record Dates: First submitted 2015-02-27; First posted 2015-03-04 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2019-12

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Hypertonic Saline; Inhaled Saline; Digestive System Diseases; Genetic Diseases, Inborn; Lung Diseases; Pancreatic Diseases; Pathologic Processes; Respiratory Tract Diseases
MeSH Terms: conditions — Cystic Fibrosis; Digestive System Diseases; Genetic Diseases, Inborn; Lung Diseases; Pancreatic Diseases; Pathologic Processes; Respiratory Tract Diseases | interventions — Saline Solution, Hypertonic; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Treatment Group (Experimental): 7% Hypertonic Saline administered via inhalation twice daily for 48 weeks
  Interventions: Drug: 7% Hypertonic Saline (HS)
- Control Group (Active Comparator): 0.9% Isotonic Saline administered via inhalation twice daily for 48 weeks
  Interventions: Drug: 0.9% Isotonic Saline (IS)

INTERVENTIONS:
Drug: 7% Hypertonic Saline (HS) — Administered via inhalation twice daily for 48 weeks. The delivery system is a PARI Sprint Junior nebulizer with a PARI Baby face mask or mouthpiece driven by a PARI Vios® compressor.
  Other Names: Hyper-Sal™, inhaled saline
  Arms: Active Treatment Group
Drug: 0.9% Isotonic Saline (IS) — Administered via inhalation twice daily for 48 weeks. The delivery system is a PARI Sprint Junior nebulizer with a PARI Baby face mask or mouthpiece driven by a PARI Vios® compressor.
  Other Names: Normal saline
  Arms: Control Group

SUMMARY:
The purpose of this study is to assess whether inhalation of 7% hypertonic saline (HS) twice daily for 48 weeks improves the lung clearance index by multiple breath nitrogen washout in comparison with inhalation of 0.9% isotonic saline (IS) in preschool children (ages 3 to 5) with cystic fibrosis.

DETAILED DESCRIPTION:
A growing body of evidence supports the importance of intervention in cystic fibrosis (CF) lung disease during early childhood, in order to potentially delay or prevent irreversible lung damage. Yet, aside from antimicrobial therapies, the CF community has no clinical trial evidence base with which to guide chronic pulmonary therapies in preschool children. Hypertonic saline (HS) is the most attractive chronic maintenance therapy to investigate in preschool children because it addresses defective mucociliary clearance, an early step in the cascade of events leading to CF lung disease that is expected to be abnormal prior to the onset of airway infection and inflammation.

Based on several studies, HS appears to be safe in children less than 6 years of age, but its effectiveness has been difficult to measure. In a previous study (ISIS), children less than 6 years old receiving HS had the same number of lung infections as children receiving a control treatment. However, the investigators think that children this young need a more sensitive test, such as lung function testing, to see if HS works in preventing lung damage. Multiple Breath Washout (MBW) is a relatively easy lung function test to perform with preschool children. It calculates a measurement called the Lung Clearance Index (LCI), a sensitive measure of airway inhomogeneity. In a sub-study of the ISIS study in 25 children, LCI improved in children that inhaled HS twice daily for 48 weeks.

This is a multicenter, randomized, double-blind, controlled, parallel group trial assessing LCI in children with CF ages 3 to 5 at enrollment. Participants will be randomized 1:1 to receive 7% HS (treatment arm) vs. 0.9 % isotonic saline (control arm) administered twice daily via jet nebulizer for 48 weeks. Study visits will occur at Screening, Enrollment, and at Weeks 12, 24, 36 and 48. Contact with a parent or legal guardian to assess adherence and interim medical history will occur at 1, 4 and 8 weeks after enrollment and then quarterly between subsequent study visits. Except for the screening visit, study visits will occur on a quarterly basis.

Total duration of participation will be up to 52 weeks. As enrollment will occur over approximately 18 months, total duration of the study is expected to be up to 30 months (18 months enrollment plus 12 months for the last participants to complete study participation).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF as evidenced by one or more clinical feature consistent with the CF phenotype or positive CF newborn screen AND one or more of the following criteria:
* A documented sweat chloride ≥ 60 milliequivalents of solute per litre (mEq/L) by quantitative pilocarpine iontophoresis (QPIT)
* A documented genotype with two disease-causing mutations in the Cystic Fibrosis Transmembrane Conductance Regulator (CFTR) gene
* Informed consent by parent or legal guardian
* Age ≥ 36 months and ≤72 months at Screening visit
* Ability to comply with medication use, study visits and study procedures as judged by the site investigator
* Ability to perform technically acceptable MBW measurements at the screening and enrollment visits

Exclusion Criteria:

* Acute intercurrent respiratory infection, defined as an increase in cough, wheezing, or respiratory rate with onset within 3 weeks preceding Screening or Enrollment visit
* Acute wheezing at Screening or Enrollment visit
* Oxygen saturation < 95% (<90% in centers located above 4000 feet elevation) at Screening or Enrollment visit
* Physical findings that would compromise the safety of the participant or the quality of the study data as determined by site investigator
* Investigational drug use within 30 days prior to Screening or Enrollment visit
* Treatment with inhaled hypertonic saline at any concentration within 30 days prior to Screening or Enrollment visit
* Chronic lung disease not related to CF
* Inability to tolerate first dose of study treatment at the Enrollment visit

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Lung Clearance Index (LCI) | 48 weeks
  Change in Lung Clearance Index (LCI) from baseline to 48 weeks measured by N2 Multiple Breath Washout (MBW) between subjects randomized to HS and IS.

SECONDARY OUTCOMES:
Change in Forced Expiratory Volume (FEV) | 48 weeks
  Change in FEV 0.75 measured by preschool spirometry between subjects randomized to HS and IS.
Pulmonary exacerbation rate | 48 weeks
  Protocol defined pulmonary exacerbation rate.
Health-related quality of life | 48 weeks
  Health-related quality of life as measured by the modified parent-reported Cystic Fibrosis Questionnaire-Revised (CFQ-R) for preschoolers.
Respiratory Signs | 48 weeks
  Parent observation of respiratory signs as measured by the Cystic Fibrosis Respiratory Sign Diary for ages 0-6 (CFRSD0-6).
Respiratory Pathogen Rate | 48 weeks
  Rates of treatment emergent CF respiratory pathogens from clinical respiratory cultures.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Davis, MD, Principal Investigator — Indiana University; Richard A Kronmal, PhD, Principal Investigator — University of Washington; Felix Ratjen, MD, PhD, FRCPC, Principal Investigator — Hospital for Sick Kids, Toronto; Margaret Rosenfeld, MD, MPH, Principal Investigator — Seattle Children's Hospital
Locations (25):
- United States (23):
  - University of Alabama-Birmingham: Pulmonary, Allergy and Critical Care Medicine, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Nemours Children's Hospital, Orlando, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children-Indiana U Med Center, Indianapolis, Indiana
  - University of Iowa, Department of Pediatrics, Iowa City, Iowa
  - Johns Hopkins University: Pediatric Pulmonary, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Women & Children's Hospital of Buffalo, Buffalo, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies Children's Hospital and Case Western Reserve University School of Medicine, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Children's Hospital of Philadelphia, UPenn, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Texas Children's Hospital and Baylor College of Medicine, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Hospital for Sick Kids, Toronto, Ontario

REFERENCES:
- [Background] Rosenfeld M, Ratjen F, Brumback L, Daniel S, Rowbotham R, McNamara S, Johnson R, Kronmal R, Davis SD; ISIS Study Group. Inhaled hypertonic saline in infants and children younger than 6 years with cystic fibrosis: the ISIS randomized controlled trial. JAMA. 2012 Jun 6;307(21):2269-77. doi: 10.1001/jama.2012.5214. PMID 22610452
- [Background] Amin R, Subbarao P, Jabar A, Balkovec S, Jensen R, Kerrigan S, Gustafsson P, Ratjen F. Hypertonic saline improves the LCI in paediatric patients with CF with normal lung function. Thorax. 2010 May;65(5):379-83. doi: 10.1136/thx.2009.125831. PMID 20435858
- [Result] Ratjen F, Davis SD, Stanojevic S, Kronmal RA, Hinckley Stukovsky KD, Jorgensen N, Rosenfeld M; SHIP Study Group. Inhaled hypertonic saline in preschool children with cystic fibrosis (SHIP): a multicentre, randomised, double-blind, placebo-controlled trial. Lancet Respir Med. 2019 Sep;7(9):802-809. doi: 10.1016/S2213-2600(19)30187-0. Epub 2019 Jun 6. PMID 31178421